CLINICAL TRIAL: NCT00192426
Title: A Prospective, Randomized, Partially-Blinded, Placebo-Controlled, Phase III, Multicenter Trial to Assess Safety, Tolerability and Immunogenicity of Liquid CAIV-T Administered Concomitantly With OPV in Healthy Children
Brief Title: Trial to Evaluate the Immune Response to OPV When Administered Concomitantly With CAIV-T to Healthy Children.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: D153-P511
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-10-03 (Estimated); Status verified 2006-10

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

INTERVENTIONS:
Biological: CAIV-T

SUMMARY:
Phase III trial to evaluate the immune response to oral poliovirus vaccine (OPV) when administered concomitantly with CAIV-T to healthy children.

ELIGIBILITY:
Inclusion Criteria:

* who are aged at least 6 months and less than 36 months of age at the time of first vaccination
* who have received a full primary vaccination schedule consisting of three doses of OPV in the first year of life
* who are in good health as determined by medical history, physical examination and clinical judgement
* whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained
* who, along with their parent(s)/legal guardian(s), will be available for duration of the trial (3 months)
* whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria:

* whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease
* with Down's syndrome or other known cytogenetic disorders
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids (see Section 4.2.1)
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study
* have an immunosuppressed or an immunocompromised individual living in the same household
* who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational)
* with a documented history of hypersensitivity to egg or egg protein or any other component of the assigned study vaccine
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to vaccination or for which use is anticipated during the study
* with any medical conditions that in the opinion of the Investigator might interfere with interpretation of the study results.

If any of these criteria are met following enrollment, the subject will be excluded from subsequent vaccine dosing.

Note: Pregnancy in a household member or any person who has regular contact with the subject is not a contraindication to the enrollment or ongoing participation of the subject in the study.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2400
Dates: Start 2001-09; Study Completion 2001-12

PRIMARY OUTCOMES:
The primary immunogenicity endpoint is the proportion of subjects achieving a post-vaccination serum antibody response for each antigen component of OPV and CAIV-T.

SECONDARY OUTCOMES:
The secondary endpoint for immunogenicity is the geometric mean titer (GMT) of serum antibody for each antigen component of OPV or the geometric mean ratio relative to the baseline titer of CAIV-T serum antibody components.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC